CLINICAL TRIAL: NCT06160908
Title: The Safety and Efficacy of Transcranial Near-infrared Light in the Treatment of Mild-Moderate Alzheimer's Disease
Brief Title: Transcranial Near-infrared Light Therapy for Mild-Moderate Alzheimer's Disease (NIR4AD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Danyang Huichuang Medical Equipment Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023162
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core phase: sham irradiation group. (Sham Comparator)
  Interventions: Device: sham NirsCure
- Core phase: Near infrared light therapy (Experimental)
  Interventions: Device: NirsCure
- Extension phase: Near infrared light therapy (Experimental): This arm includes participants who finish the core phase from the core phase experimental group and the core phase sham comparator group. The intervention is the same as the intervention in the core phase.
  Interventions: Device: NirsCure

INTERVENTIONS:
Device: NirsCure — True near-infrared light； Once a day, once for 30 minutes, 6 times a week
  Arms: Core phase: Near infrared light therapy
Device: sham NirsCure — Non near-infrared light irradiation；only the equipment appearance is consistent with the test device；Once a day, once for 30 minutes, 6 times a week
  Arms: Core phase: sham irradiation group.
Device: NirsCure — True near-infrared light； Once a day, once for 30 minutes, 6 times a week
  Arms: Extension phase: Near infrared light therapy

SUMMARY:
The goal of this study is to explore the efficacy and safety of Near-infrared light Photobiomodulation in patients with mild-moderate Alzheimer's disease(AD).

This study will employ a randomized, double-blind, sham-controlled approach. This trial contains core phase and extension phase. In the core phase, qualified subjects were selected and randomized (experimental group: control group=1:1). The subjects who entered the experimental group received 30 minutes of near-infrared light therapy once a day, 6 times a week, for 16 weeks of continuous treatment. The subjects who entered the control group received 30 minutes of non-near-infrared light irradiation once a day (false treatment), 6 times a week, for 16 weeks. After finishing the core phase, patients from both groups of the core phase are eligible to enter the extension phase. In the extension phase, all the participants receive active near-infrared light therapy until week 196.

ELIGIBILITY:
Inclusion Criteria:

1. 50 - 90 years old, no gender limitation;
2. Meeting clinical diagnostic criteria of probable AD according to National Institute on Aging and the Alzheimer's Association (NIA-AA) guidelines;
3. Clinical Dementia Rating Scale Total Score (CDR-GS) score ≥ 1 and ≤ 2, Clinical Dementia Rating Scale Memory Box score ≥ 0.5;
4. Amyloid PET or cerebrospinal fluid examination or blood biomarkers conforms to changes in AD biomarkers;
5. The MMSE score is ≥ 12 and ≤ 26;
6. Education level is non illiterate or has received cultural education for 4-6 years or more;
7. If taking mental or cognitive improvement drugs, the dosage must be stable for at least 3 months before the study, and remain unchanged during the light regulation intervention period. Unless otherwise specified, participants must consistently use all other (i.e. non Alzheimer's disease related) permitted concomitant medications for at least 4 weeks before baseline;
8. Having a designated guardian or caregiver who can assist them in participating in the experiment (defined as someone who can support participants throughout the entire study period and spend at least 8 hours with them per week);
9. Subjects with informed consent;

Exclusion Criteria:

1. Any neurological and psychiatric symptoms beyond the scope of symptoms that can be caused by Alzheimer's disease;
2. A history of transient ischemic attack (TIA), stroke, or epilepsy within 12 months;
3. Any mental diagnosis or symptoms that may interfere with the participant's research process (such as hallucinations, severe depression, or delusions);
4. Contraindications to MRI, including pacemakers/defibrillators, ferromagnetic metal implants, etc;
5. MRI shows other clinically significant lesions, which may indicate the diagnosis of dementia beyond Alzheimer's disease;
6. MRI shows other important pathological findings, including but not limited to: 4 or more microbleeds with a diameter of 10 millimeters or less; Single bleeding lesion with a maximum diameter greater than 10 millimeters; Surface iron deposition area; Evidence of exudative edema; Evidence of brain contusion, encephalomalacia, aneurysm, vascular malformation, or infectious disease; Multiple lacunar infarcts or strokes involving major vascular areas, severe small vessel or white matter lesions; Space occupying lesions; Or brain tumors (diagnosed as meningiomas or arachnoid cysts, lesions with a maximum diameter of less than 1 cm may not be ruled out);
7. A photosensitive response to sunlight or visible light, with eczema or increased sensitivity on the skin at the intervention site;
8. Severe visual or hearing impairment;
9. Individuals who are addicted to alcohol, drugs, or other drugs or have a tendency to become addicted;
10. Participating in other AD clinical trials;
11. Any other medical conditions that are not stable and adequately controlled (such as heart, respiratory, gastrointestinal, kidney diseases), or situations that the researcher believes may affect the safety of participants or interfere with the evaluation of the study;
12. Other conditions that, in the opinion of the investigator, may not be suitable for this study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline on the Alzheimer's disease assessment scale-cognitive section(ADAS-Cog) | 16 weeks

SECONDARY OUTCOMES:
change from baseline on the Alzheimer's disease assessment scale-cognitive section(ADAS-Cog) | baseline, 8 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
change from baseline on the Mini Mental state Examination (MMSE) score | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
change from baseline on the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
change from baseline on the Alzheimer's Disease Cooperative study-clinical global impression of change scale(ADCS-CGIC) | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
change from baseline on the Alzheimer's Disease Cooperative study-Activities of Daily Living Scale(ADCS-ADL) | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
change from baseline on the Neuropaychiatic Inventory (NPI) | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
change from baseline on the Hamilton depression scale (HAMD) | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
Change from Baseline in Brain Amyloid Plaque Deposition as measured by PET Scan | baseline,16 weeks, 52 weeks, 76 weeks, 100 weeks, 148 weeks, 196 weeks.
Change from Baseline in FDG-PET imaging | baseline,16 weeks, 52 weeks, 76 weeks, 100 weeks, 148 weeks, 196 weeks.
Change from Baseline in resting state Electroencephalogram and Event Related Potentials (ERP) | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
Change from Baseline in resting state near-infrared brain function imaging | baseline,8 weeks,16 weeks, 28 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks.
Change from Baseline in magnetic resonance imaging analysis | baseline, 8 weeks,16 weeks, 40 weeks, 52 weeks, 64 weeks, 76 weeks, 88 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.
Change from baseline in blood biomarkers. | baseline, 8 weeks,16 weeks, 52 weeks, 76 weeks, 100 weeks, 124 weeks, 148 weeks, 172 weeks, 196 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, MD., PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No